CLINICAL TRIAL: NCT03731585
Title: Online Psychosocial Intervention for Women With Lung Cancer Undergoing Treatment
Brief Title: Online Psychosocial Intervention in Improving Social Well-Being and Support in Women With Stage I-IV Non-small Cell Lung Cancer Undergoing Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0501; NCI-2018-02113 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0501 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-10-12; First posted 2018-11-06 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Behavior Therapy; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (psychological intervention) (Experimental): Patients participate in 5 psychological sessions and complete training on mindfulness, compassion, emotional processing, social support, generating positive emotions, and proactive coping strategies once a week for up to 5 weeks. Patients also complete questionnaires over 35 minutes and participate in video-based group sessions weekly for 5 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Questionnaire Administration; Procedure: Support Group Therapy
- Group II (educational intervention) (Experimental): Patients participate in 5 information sessions and receive education on lung cancer, symptom management, communication, and practicing self-care once a week for up to 5 weeks. Patients also complete questionnaires and participate in group sessions as in group I.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration; Procedure: Support Group Therapy

INTERVENTIONS:
Behavioral: Behavioral Intervention — Participate in psychological sessions
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Group I (psychological intervention)
Other: Educational Intervention — Participate in educational sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (educational intervention)
Other: Questionnaire Administration — Ancillary studies
Procedure: Support Group Therapy — Participate in group sessions

SUMMARY:
This trial studies how well online psychosocial intervention works in improving social well-being and support in women who are undergoing treatment for stage I-IV non-small cell lung cancer. Psychosocial intervention techniques, such as mindfulness, compassion, and emotional processing, may improve distress and help patients manage symptoms related to non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the feasibility (primary outcome) of the BREATHE intervention in women with lung cancer (LC).

SECONDARY OBJECTIVES:

I. Establish the initial intervention efficacy regarding psychological distress (secondary outcome) and cancer symptoms (tertiary outcome) relative to an education comparison (EC) group.

EXPLORATORY OBJECTIVES:

I. Explore potential mediation (e.g., mindfulness, compassion, inflammatory processes) and moderation (e.g., demographic and medical factors) of the intervention effects.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (PSYCHOLOGICAL): Patients participate in 5 psychological sessions and complete training on mindfulness, compassion, emotional processing, social support, generating positive emotions, and proactive coping strategies once a week for up to 5 weeks. Patients also complete questionnaires over 35 minutes and participate in video-based group sessions weekly for 5 weeks.

GROUP II (EDUCATIONAL): Patients participate in 5 information sessions and receive education on lung cancer, symptom management, communication, and practicing self-care once a week for up to 5 weeks. Patients also complete questionnaires and participate in group sessions as in group I.

After completion of study intervention, patients are followed up at 1 week and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with stage I-IV non-small cell lung cancer within 3 months of diagnosis at the time of recruitment and receiving any type of treatment at the time of recruitment. For women with metastatic disease, disease must be stable (without disease progression based on patients' latest imaging impressions) per treating oncologist
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Have access to the internet
* Able to read, write and speak English

Exclusion Criteria:

* Major psychiatric or cognitive deficits that would impede the completion of self-report instruments as deemed by the clinical team
* Regular (self-defined) participation in psychotherapy or a formal cancer support group

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
BREATHE intervention in women with Lung Cancer determined successful by overall accrual | Up to 3 months
  Overall accrual assessed by ≥ 50% of eligible patients consent (i.e., approach 140 to achieve 70 that consent).
BREATHE intervention in women with Lung Cancer determined successful by attrition | Up to 3 months
  Attrition assessed by ≥ 71% of enrolled patients (≥ 50 patients) complete T1 and T2 assessments;
BREATHE intervention in women with Lung Cancer determined successful by adherence | Up to 3 months
  Adherence assessed by ≥ 75% of all practice sessions are attended in each arm.
BREATHE intervention in women with Lung Cancer determined successful by acceptability | Up to 3 months
  Acceptability assessed by ≥ 75% of participants indicating that the program is useful and enjoyable in each arm.

SECONDARY OUTCOMES:
Efficacy regarding psychological distress: CES-D | Up to 3 months
  The study will examine preliminary evidence of intervention efficacy. Will calculate effect sizes for between-group comparisons based on the primary efficacy endpoint of Center for Epidemiologic Studies Depression Scale (CES-D), a 20-item self-report measure focusing on the affective component of depression.
  Answers range from: almost never (less than 1 day), sometimes (1 to 2 days), often (3 to 4 days), almost always (5 to 7 days).
Efficacy regarding cancer symptoms: IES | Up to 3 months
  The study will examine preliminary evidence of intervention efficacy. Will calculate effect sizes for between-group comparisons based on the primary efficacy endpoint of Impact of Event Scale (IES) measured at T2 using analysis of covariance (ANCOVA). IES scale answers range from NOT AT ALL, RARELY, SOMETIMES, OFTEN.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Milbury K, Kroll J, Chen A, Antonoff MB, Snyder S, Higgins H, Yang CC, Li Y, Bruera E. Pilot Randomized Controlled Trial in Women With Non-Small Cell Lung Cancer to Assess the Feasibility of Delivering Group-Based Psychosocial Care via Videoconference. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211052520. doi: 10.1177/15347354211052520. PMID 34663123
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org